CLINICAL TRIAL: NCT05833620
Title: Identification and Functional Characterization of Genetic Variants Associated With Specific Clinical Phenotypes in Hereditary Angioedema Due to C1 Inhibitor Deficiency: An Unbiased Approach
Brief Title: Identification and Characterization of Genetic Variants in Hereditary Angioedema
Acronym: GENOMAEH_01
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: GENOMAEH_01
Record Dates: First submitted 2023-03-17; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hereditary Angioedema With C1 Esterase Inhibitor Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic patients: Adult patients (≥ 18 years old) with hereditary angioedema with C1INH deficiency (HAE-C1INH) from different regions of Spain will be included. Patients included in the study will be divided into two groups: a) symptomatic, which will be those who present symptoms compatible with HAE-C1INH and who have a confirmed diagnosis
- Asymptomatic patients: Asymptomatic patients, which will be those with a C1INH deficiency and who have not developed symptoms of HAE. Asymptomatic patients must be at least 22 years old and meet the same criteria than those symptomatic, except for the presence of symptoms consistent with HAE-C1INH

SUMMARY:
This project aims to analyse in an unbiased way the existence of genetic variants that contribute to explaining and predicting the differences in clinical expression between patients with HAE.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) with HAE-C1INH diagnosis (confirmed by mutation in SERPING1 gen or immunochemical study showing a decrease in C1INH function <50% in two determinations together with a family history (symptomatic patients' group)
* Patients ≥ 22 years old with C1INH hereditary deficiency (confirmed by mutation of SERPING1 gene or immunochemical study showing a decrease in C1INH function <50% in two determinations together with a family history) and who have not developed symptoms consistent with HAE-C1INH
* Signed informed consent.

Exclusion Criteria:

* No confirmed C1INH deficiency.
* Inability to sign the informed consent.
* Presence of recurrent angioedema with histaminergic characteristics (response to treatment with antihistamines, glucocorticoids and/or epinephrine)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with hereditary angioedema with C1INH deficiency (HAE-C1INH) from different regions of Spain will be included. Patients included in the study will be divided into two groups: a) symptomatic (≥ 18 years old), which will be those who present symptoms compatible with HAE-C1INH and who have a confirmed diagnosis and b) asymptomatic patients (≥ 22 years old), which will be those with a C1INH deficiency and who have not developed symptoms of HAE.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Set of validated disease-modifying genetic variants in Spanish patients with HAE-C1INH | Day 1
  To identify and characterize novel genetic variants associated with the incomplete penetrance and variable clinical expressivity observed in HAE-C1INH patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No